CLINICAL TRIAL: NCT01376804
Title: Tolerability of up to 200 Days of Valganciclovir Oral Solution or Tablets in Pediatric Kidney Transplant Recipients
Brief Title: A Study of Oral Valcyte (Valganciclovir) in Pediatric Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NV25409; 2010-022514-47 (EudraCT Number)
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Kidney Transplantation, Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valganciclovir (Experimental): Participants received a once daily oral dose (solution or tablets) of valganciclovir starting within 10 days of kidney transplant for up to 200 days post-transplant. Dose (in milligrams) was calculated using the algorithm [7 * Body Surface Area * Creatinine Clearance].
  Interventions: Drug: valganciclovir [Valcyte]

INTERVENTIONS:
Drug: valganciclovir [Valcyte] — Oral, daily for up to 200 days.

SUMMARY:
This open-label, single arm study will evaluate the tolerability and efficacy of Valcyte (valganciclovir) in the prevention of cytomegalovirus disease in pediatric renal transplant recipients. After transplantation, patients (aged 4 months to 16 years) will receive Valcyte orally daily for up to 200 days post-transplant and will be followed for 52 weeks post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Children, 4 months to 16 years of age
* Patient has received a kidney transplant
* At risk of developing cytomegalovirus disease
* Adequate hematological and renal function
* Able to tolerate oral medication
* Negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* Allergic or significant adverse reaction to acyclovir, valacyclovir or ganciclovir in the past
* Severe uncontrolled diarrhea (more than 5 watery stools per day)
* Liver enzyme elevation of more than five times the upper limit of normal for aspartate aminotransferase [AST (SGOT)] or alanine aminotransferase [ALT (SGPT)]
* Patient requires use of any protocol prohibited concomitant medication
* Previous participation in this clinical study

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2011-07-31 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (4):
  - University of Florida Pediatric Nephrology, Gainesville, Florida
  - UCLA Center For Health Sciences; Division of Pediatric Nephrology, Los Angeles, Louisiana
  - Mount Sinai Medical Center, New York, New York
  - Uni of Utah Health Science Center; Pediatric Nephrology, Salt Lake City, Utah
- Australia (3):
  - Children'S Hospital At Westmead; Department of Nephrology, Westmead, New South Wales
  - Mater Childrens Hospital, South Brisbane, Herston, Queensland
  - Royal Children'S Hospital; Department of Nephrology, Parkville, Victoria
- Universidade Federal de Sao Paulo - UNIFESP, São Paulo, São Paulo, Brazil
- France (3):
  - CHU de Nantes - Service de pédiatrie, Nantes
  - Hôpital Robert Debré; Nephrologie pediatrique, Paris
  - Hop Necker Enfants Malades;Nephrologie Pediatrique, Paris
- Germany (4):
  - Klinik und Poliklinik für Kinder- und Jugendmedizin- Köln, Uniklinik Köln, Cologne
  - Universitätsklinikum für Kinder und Jugendmedizin Hamburg, Hamburg
  - KfH Nierenzentrum für Kinder und Jugendliche an der MHH Hannover, Hanover
  - Klinik Kinderheikunde I des Zentrums für Kinder- und Jugendmedizin, Universität Heidelberg, Heidelberg
- Mexico (3):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Instituto Mexicano de Transplantes, Cuernavaca
  - Hospital Infantil de Mexico Federico Gomez, México
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz: Nefrologia Pediatrica, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Nefrologia Pediatrica, Seville
- Sahlgrenska Sjukhuset; Transplantationskirurgiska Kliniken, Gothenburg, Sweden
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital For Children, Bristol
  - Royal Hospital For Sick Children; Dept. of Child Health, Glasgow

RESULTS

PARTICIPANT FLOW:
Groups:
- Valganciclovir: Participants received a once daily oral dose (solution or tablets) of valganciclovir starting within 10 days of kidney transplant for up to 200 days post-transplant. Dose [in milligrams (mg)] was calculated using the algorithm [7 * Body Surface Area * Creatinine Clearance].
Period: Treatment Period
Arm/Group | Valganciclovir
Started | 57
Received Study Drug | 56
Completed | 49
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 6
Not completed — Patient did not receive study drug | 1
Period: Follow-up Period
Arm/Group | Valganciclovir
Started | 55 (6 of the 7 patients who withdrew from treatment continued to the Follow-up Period.)
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures were based on the Intent-to-treat population that included all enrolled patients who had taken at least one dose of study drug.
Groups:
- Valganciclovir: Participants received a once daily oral dose (solution or tablets) of valganciclovir starting within 10 days of kidney transplant for up to 200 days post-transplant. Dose (in mg) was calculated using the algorithm [7 * Body Surface Area * Creatinine Clearance].
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Age, Customized [Number; unit: Participants]
  ≤ 2 Years | 6 (0.5)
  > 2 to < 12 Years | 18 (2.5)
  ≥ 12 Years | 32 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE) or Withdrawal Due to AEs
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. Pre-existing conditions which worsen during a study were reported as AEs.
  A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: 52 weeks
Population: Safety Population included all enrolled patients who received at least one dose of study medication and had at least one post-baseline assessment of safety.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants
  Adverse Events | 56
  Serious Adverse Events | 41
  Withdrawals due to AE | 6

2. Secondary Outcome: Number of Participants With Cytomegalovirus (CMV) Infection in the First 52 Weeks Post-Transplant as Assessed by the Investigator
Description: A polymerase chain reaction (PCR) based assay or antigenaemia assay was used for the qualitative assessment of CMV viremia (presence of CMV in the blood) by each study center as part of the clinical assessment required for diagnosis of CMV infection.
Time Frame: 52 weeks
Population: Intent-to-treat (ITT) population included all enrolled patients who had taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants | 3

3. Secondary Outcome: Number of Participants With Cytomegalovirus (CMV) Disease in the First 52 Weeks Post-Transplant as Assessed by the Investigator
Description: A polymerase chain reaction (PCR) based assay or antigenaemia assay was used for the qualitative assessment of CMV viremia by each study center as part of the clinical assessment required for diagnosis of CMV infection. CMV disease included CMV syndrome or tissue invasive CMV. CMV syndrome required fever ≥ 38 degrees Celsius, severe malaise, leukopenia on 2 separate measurements, atypical lymphocytosis ≥ 5%, thrombocytopenia, elevation of hepatic transaminases and presence of CMV in blood. Tissue Invasive CMV required evidence of localized CMV infection in a biopsy or other appropriate symptom and relevant symptoms or signs of organ dysfunction.
Time Frame: 52 weeks
Population: Intent-to-treat (ITT) population included all enrolled patients who had taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants
  CMV Syndrome | 1
  Tissue Invasive CMV | 0

4. Secondary Outcome: Number of Participants With Peak Cytomegalovirus (CMV) Viral Load up to Week 52 Post-Transplant
Description: Blood samples were sent to a central lab for the quantitative assessment of CMV viral load (amount of CMV in the blood) by an FDA-approved molecular-based assay. The number of participants in each category is reported in copies/milliliter (CP/mL). CMV DNA is detected in all categories < 150 CP/mL and above.
Time Frame: 52 weeks
Population: ITT population included all enrolled patients who had taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants
  No CMV DNA Detected | 30
  < 150 CP/mL | 16
  150 to 1,000 CP/mL | 6
  1,001 to 5,000 CP/mL | 3
  > 5,000 CP/mL | 1

5. Secondary Outcome: Number of Participants With Biopsy Proven Rejection
Description: Renal biopsies were performed as medically indicated. Biopsies were assessed histologically using the updated Banff criteria 1997.
Time Frame: 52 Weeks
Population: ITT population included all enrolled patients who had taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants
  ≤ 2 Years | 1
  >2 to <12 Years | 1
  ≥ 12 Years | 3

6. Secondary Outcome: Number of Participants With Graft Loss
Description: Graft loss was defined as the institution of chronic dialysis (at least 6 consecutive weeks), transplant nephrectomy, or retransplantation.
Time Frame: 52 Weeks
Population: ITT population included all enrolled patients who had taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants | 0

7. Secondary Outcome: Number of Participants With Death
Time Frame: 52 Weeks
Population: ITT population included all enrolled patients who had taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 56
Participants | 0

8. Secondary Outcome: Number of Participants With Known Ganciclovir Resistance (Mutations in Either UL54 or UL97 Genes)
Description: All patients with measurable CMV had both UL54 and UL97 genes sequenced to assess for known CMV resistance to ganciclovir.
Time Frame: 52 Weeks
Population: All patients meeting the resistance analysis criteria are included into the resistance analysis.
Measure: Number; unit: Participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 10
Participants
  UL54 | 0
  UL97 | 1

ADVERSE EVENTS:
Arm/Group | Valganciclovir
Serious Adverse Events (participants affected / at risk) | 41/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir (N=56)
Urinary Tract Infection (Infections and infestations) | 7
Escherichia Urinary Tract Infection (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 4
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3
Bacterial Pyelonephritis (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Viral Infection (Infections and infestations) | 2
Chronic Sinusitis (Infections and infestations) | 1
Diarrhoea Infectious (Infections and infestations) | 1
Gastroenteritis Norovirus (Infections and infestations) | 1
Gastrointestinal Protozoal Infection (Infections and infestations) | 1
Gastrointestinal Viral Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia Mycoplasmal (Infections and infestations) | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 1
Rotavirus Infection (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Urinary Tract Infection Bacterial (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Bicytopenia (Blood and lymphatic system disorders) | 1
Bladder Dysfunction (Renal and urinary disorders) | 1
Neurogenic Bladder (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Ureteric Obstruction (Renal and urinary disorders) | 1
Urethral Obstruction (Renal and urinary disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Vesicoureteric Reflux (Renal and urinary disorders) | 1
Blood Creatinine Increased (Investigations) | 5
HLA Marker Study Positive (Investigations) | 1
Transplant Rejection (Immune system disorders) | 3
Kidney Transplant Rejection (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Complications Of Transplant Surgery (Injury, poisoning and procedural complications) | 1
Complications Of Transplanted Kidney (Injury, poisoning and procedural complications) | 1
Benign Intracranial Hypertension (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Papilloedema (Eye disorders) | 1
Device Leakage (General disorders) | 1
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Vesicoureteral Reflux Surgery (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir (N=56)
Upper respiratory tract infection (Infections and infestations) | 20
Urinary tract infection (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 6
BK virus infection (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 4
Escherichia urinary tract infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Leukopenia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 12
Anaemia (Blood and lymphatic system disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 18
Abdominal pain (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 12
Tremor (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 3
Dysuria (Renal and urinary disorders) | 10
Haematuria (Renal and urinary disorders) | 6
Renal tubular acidosis (Renal and urinary disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 3
Blood creatinine increased (Investigations) | 7
Weight increased (Investigations) | 4
Pyrexia (General disorders) | 9
Oedema peripheral (General disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 3
Insomnia (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.